CLINICAL TRIAL: NCT04531358
Title: Demonstration of an Anti-allergic Effect in Subjects Treated With Callergin Nasal Spray in Comparison to Untreated Subjects and Subjects Treated With Vis Alpin® Alpensalz Nasal Spray, All Suffering From Grass Pollen Induced Rhinitis/Rhinoconjunctivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marinomed Biotech AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAL_19_01
Record Dates: First submitted 2020-08-21; First posted 2020-08-28 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-10

CONDITIONS: Allergic Rhinitis; Allergic Rhinoconjunctivitis
Keywords: Allergic Rhinoconjunctivitis; Allergic Rhinitis; Callergin; Vienna Challenge Chamber; Total Nasal Symptom Score; Carrageenan; Carragelose; Iota-carrageenan
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, double-blinded randomized three-way cross-over single site study In the cross-over setting two treatments, namely Callergin and Vis Alpin® Alpensalz will be evaluated compared to untreated subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Callergin (Active Comparator): One puff (140 microliter) into each nostril
  Interventions: Device: nasal spray
- Alpin Alpensalz (Active Comparator): One puff (140 microliter) into each nostril
  Interventions: Device: nasal spray
- no treatment (Experimental): Patients do not receive a treatment
  Interventions: Other: no treatment

INTERVENTIONS:
Device: nasal spray — application of nasal spray
  Arms: Alpin Alpensalz; Callergin
Other: no treatment — no treatment
  Arms: no treatment

SUMMARY:
Allergic rhinitis (AR) in its seasonal and perennial form is a common allergic condition. The majority of allergic rhinitis sufferers report nasal (congestion, sneezing, itching and rhinorrhea) and ocular (redness, watery eyes, itching and burning) symptoms.

The polymer Carragelose® is a unique broadly active anti-viral compound for treating respiratory diseases. Carragelose® is a sulfated polymer from red seaweed also widely used in the food industry and has GRAS status (FDA). The compound has a broad spectrum of anti-viral properties. Sprayed into the nose Carragelose® creates a protective layer in the nasal cavity which could prevent allergic rhinitis symptoms as well. This anti-allergic clinical performance compared to untreated subjects and to subjects treated with Vis Alpin® Alpensalz nasal spray should be demonstrated.

No clinical data in humans have been generated with Callergin so far. Callergin nasal spray is a certified Class I medical device. The use of the nasal spray is associated with a very low risk for patients. Callergin is used to moisturize nasal mucosa and to support the treatment of rhinitis of any kind. Allergic subjects could benefit from the moisturizing protective layer on the nasal mucosa, which could prevent allergen attachment to the mucosa surface.

This will be a prospective, controlled, double-blinded randomized three-way cross-over single site study in adult subjects (18 to 65 years) who demonstrate a grass pollen specific Immunoglobulin E (IgE) reactivity and have a history of grass pollen induced allergic rhinitis/rhinoconjunctivitis with or without controlled asthma. In the cross-over setting two treatments, namely Callergin and Vis Alpin® Alpensalz will be evaluated compared to untreated subjects. The subjects will be treated with one puff (140 microliter) into each nostril.

The primary objective of the trial is to demonstrate an anti-allergic clinical performance of Callergin nasal spray compared to untreated subjects in grass pollen induced rhinitis/rhinoconjunctivitis. The evaluation will be based on the assessment of rhinitis symptoms during grass pollen challenge performed in the Vienna Challenge Chamber (environmental exposure chamber).

Secondary objective of the trial is to demonstrate an anti-allergic clinical performance of Callergin nasal spray compared to subjects treated with Vis Alpin® Alpensalz nasal spray.

DETAILED DESCRIPTION:
This is a prospective, controlled, double-blinded randomized three-way cross-over single site study in adult subjects (18 to 65 years) who demonstrate a grass pollen specific Immunoglobulin E (IgE) reactivity and have a history of grass pollen induced allergic rhinitis/rhinoconjunctivitis with or without controlled asthma. In the cross-over setting two treatments, namely Callergin and Vis Alpin® Alpensalz will be evaluated compared to untreated subjects.

Visit 1 - Screening:

At least one week prior to first treatment block, subjects will be screened for appropriate allergic response. A total nasal symptom score (TNSS) of at least 6 points out of 12 within the first two hours in the grass pollen challenge chamber is required to be included into the study. If a screening for appropriate allergic response was done during the last 12 months, results from this allergy challenge can be used to fulfil the respective inclusion criteria.

Visit 2 - Inclusion:

In addition to the screening provocation the medical and allergic history, safety lab as well as retrieving inclusion and exclusion criteria will be assessed via anamnesis. Furthermore, all safety assessments will be conducted.

Note: Visit 1 and visit 2 could be done on the same day!

Visit 3: Day1 of first treatment period Eligible subjects will be randomly assigned to one of the two treatment arms (fully blinded) and to the untreated control group in the order of appearance and their screening numbers assigned at visit 1. Subjects will enter the study site about one hour ahead of the start of allergen provocation. After positive completion of all study relevant assessments, subjects will be randomized and handed out their specific nasal spray. Ten to five minutes ahead of entering the grass pollen challenge chamber the treatment (nasal spray) application in the two treatment groups will take place under staff supervision. Afterwards the chamber session starts for subjective and objective assessments for a period of 3 hours.

The subjective nasal symptom score will be recorded every fifteen minutes during a 3-hour allergen exposure challenge. Every hour rhinomanometry will be performed to objectively evaluate blockage of the nose. An additional rhinomanometry will be performed 30 minutes after entry.

Visit 4: Day1 of second treatment period Subjects will enter the study site about one hour ahead of the start of allergen provocation. According to randomization number, subjects in the two treatment groups will receive the respective nasal spray. In the following Visit 4 will be done in the same way as Visit 3.

Visit 5: Day1 of third treatment period Subjects will enter the study site about one hour ahead of the start of allergen provocation. According to randomization number, subjects in the two treatment groups will receive the respective nasal spray. In the following Visit 5 will be done in the same way as Visit 3.

Between the respective study treatments, a wash-out period of at least 7 days must be adhered to allowing complete symptom relief from previous challenge. After the wash-out period, subjects change to the next treatment block in the sequence.

During the entire trial, subjects will be asked to monitor for adverse events (AEs), and they will record the use of concomitant medications on the provided form.

One week after the final provocation session, subjects will complete the trial after their follow up visit.

The trial design is appropriate for the indication studied. Validated methods of data collection, analysis, and evaluation will be used for the trial.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before any trial related procedures are performed
* Healthy male or female subjects aged 18 to 65 years
* A documented clinically relevant allergic history of moderate to severe SAR to grass pollen for the previous two years
* Subjects exhibit a moderate to severe response to approximately 1500 grass pollen grains/m3 within the first 2 hours in the Vienna Challenge Chamber, which is defined as total nasal symptom score (TNSS) of at least 6 (out of 12) using standard VCC grass pollen allergen mixture. Nasal symptom score is the sum of "nasal congestion", "rhinorrhea", "itchy nose" and "sneezing", each of which have been scored on a categorical scale from 0 to 3.
* Positive Skin Prick Test (SPT) response (wheal diameter at least 3 mm larger than diluent control) to grass pollen SPT solutions (standard Allergopharma) at screening or within the last 12 months prior to study start.
* Positive serum specific IgE against recombinant major allergen components of the used grass pollen e.g. g6 (specific CAP IgE ≥0.70 kU/L) at screening or within the last 12 months prior to study start.
* Asthma patients only if the asthma condition is mild or intermittent, and if those are not treated with steroids
* Subject has a forced expiratory volume in 1 second (FEV1) of at least 80% of predicted value (ECCS) at the screening.
* Subject is capable of understanding the study procedures and potential risks associated with the study, and voluntarily agrees to participate by giving written informed consent.
* Subject is able to adhere to dose and visit schedules.
* Subject is able to read, understand and

Exclusion Criteria:

* A clinical history of uncontrolled asthma within 3 months prior to screening
* Subjects with asthma requiring treatment with inhaled corticosteroids on a regular basis judged by the investigator
* Previous successful immunotherapy to grass pollen, a grass pollen allergen or a cross-reacting allergen within the past 3 years
* Ongoing treatment with any allergen-specific immunotherapy product
* Subjects with history of tuberculosis
* Symptoms of or treatment for upper respiratory tract infection, acute sinusitis, acute otitis media or other relevant infectious process at randomization
* Clinically relevant nasal polyps, medical history of paranasal sinus surgery and/or medical history of surgery of nasal turbinates judged by the investigator
* Subjects using any ophthalmic steroids during the last 30 days
* Subjects treated with nasal, inhaled or systemic steroids during the last 30 days
* History of anaphylaxis with cardiorespiratory symptoms (immunotherapy, exercise induced, food allergy, drugs or an idiopathic reaction)
* Any clinically relevant chronic disease judged by the investigator
* Systemic disease affecting the immune system judged by the investigator
* Use of an investigational drug within 30 days/5 half-lives of the drug (which ever longest) prior to screening
* History of allergy, hypersensitivity or intolerance to any ingredients of the study medication
* History of alcohol or drug abuse.
* Being immediate family of the investigator or trial staff, defined as the investigator's/staff's spouse, parent, child, grandparent or grandchild
* Subjects treated with leukotriene antagonists (1 month before study start), long- lasting anti-histamines, like cetirizine, fexofenadine, loratadine, desloratadine, hydroxyzine (5 to 10 days before study start), mast cell stabilizer (2 weeks before study start) or nasal decongestant (3 days before study start)
* Subjects with an acute or chronic sinusitis judged by the investigator
* Positive Serology result judged by the investigator
* Pregnant, lactating or sexually active women with childbearing potential who are not using a medically accepted and s

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | 0-3 hours of grass pollen allergen exposure challenge
  The TNSS is the sum of the four individual symptoms
  * nasal congestion
  * rhinorrhoea
  * itchy nose
  * sneezing each scored on a 4-point categorical scale from 0-3 with "0"= none "1"=mild "2"=moderate "3"=severe

SECONDARY OUTCOMES:
Nasal airflow | 0-3 hours of grass pollen allergen exposure challenge
  Anterior nasal airflow will be assessed by rhinomanometry.
Nasal secretion | 0-3 hours of grass pollen allergen exposure challenge
  Tissue weights will be used to assess nasal secretion
Total ocular symptom score (TOSS) | 0-3 hours of grass pollen allergen exposure challenge
  Total ocular symptom score (TOSS) is the sum of the symptoms "ocular itching", "redness", "watery eyes".
  Each individual symptom of TOSS will be scored on a 4-point categorical scale from 0-3 (where "0"= none "1"=mild "2"=moderate "3"=severe). TOSS will be assessed every 15 minutes during the three hours grass pollen allergen exposure challenge.
Total asthma symptom score (TASS) | 0-3 hours of grass pollen allergen exposure challenge
  Total asthma symptom score (TASS) is the sum of the symptoms "cough", "wheeze", "dyspnea".
  Each individual symptom of TASS will be scored on a 4-point categorical scale from 0-3 (where "0"= none "1"=mild "2"=moderate "3"=severe). TASS will be assessed every 15 minutes during the three hours grass pollen allergen exposure challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Prieschl-Grassauer, PhD, Study Chair — CSO
Locations (1):
- Ordination Dr. Petra Zieglmayer Vienna Challenge Chamber, Vienna, Austria

REFERENCES:
- [Derived] Unger-Manhart N, Morokutti-Kurz M, Zieglmayer PU, Lemell P, Savli M, Zieglmayer R, Prieschl-Grassauer E. Carrageenan-Containing Nasal Spray Alleviates Allergic Symptoms in Participants with Grass Pollen Allergy: A Randomized, Controlled, Crossover Clinical Trial. Int J Gen Med. 2024 Feb 3;17:419-428. doi: 10.2147/IJGM.S447359. eCollection 2024. PMID 38333020